CLINICAL TRIAL: NCT00880555
Title: Semantic Memory, Financial Capacity and Brain Perfusion in MCI
Brief Title: Semantic Memory, Financial Capacity, and Brain Perfusion in Mild Cognitive Impairment (MCI) (CASL)
Acronym: CASL
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: E6553-W
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Magnetic Resonance Imaging; Alzheimer disease; Mild cognitive impairment; Continuous arterial spin labeling; Semantic memory
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — N/A- no biospecimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Arm 1: Non-Dementia Memory Disorder: Elderly patients with non-dementia memory disorder (mild cognitive impairment)
- Arm 2: Control: Elderly controls without memory impairment
- Arm 3: Mild Alzheimer Disease: Patients with mild Alzheimer disease (but preserved routine activities of daily living)

SUMMARY:
Alzheimer's disease (AD) often manifests as a memory disorder before dementia develops. Dementia is considered to be present when a person can no longer handle complex activities of daily living, such as managing finances. This study will investigate the relationship between changes in the ability to manage finances and brain perfusion, which will be measured using continuous arterial spin-labeling (an experimental MRI). Subjects will also undergo neuropsychological tests focusing on several types of memory and thought process, with special emphasis on semantic memory. An important question to be addressed is whether changes in function are better predicted by the neuropsychological tests or by the brain scan.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) often manifests as a memory disorder before dementia develops. Dementia is considered to be present when a person can no longer handle complex activities of daily living, such as managing finances. This study will investigate the relationship between changes in the ability to manage finances and brain perfusion, which will be measured using continuous arterial spin-labeling (an experimental MRI). Subjects will also undergo neuropsychological tests focusing on several types of memory and thought process, with special emphasis on semantic memory. An important question to be addressed is whether changes in function are better predicted by the neuropsychological tests or by the brain scan. Participants will undergo a single MRI scan, baseline financial capacity instrument (FCI) and cognitive evaluation, and then will be followed approximately annually to repeat the functional and cognitive assessments. Linear mixed effects models will be used to fit a model predicting financial capacity based on baseline cognitive tests. Measures from the MRI scan will be added to the model to determine whether imaging improves the predictions.

ELIGIBILITY:
Inclusion Criteria:

* Veteran or non-veteran
* Age 50-89
* With normal cognition or memory impairment (MCI or mild AD)
* English speaking
* Right handed
* Adequate vision and hearing to take part in tests
* Able and willing to undergo MRI scan
* Medically and psychiatrically stable
* No other brain disease (such as tumor, Parkinson's disease, major stroke)

Exclusion Criteria:

* Pregnancy
* Inability to tolerate MRI (due to metal in body or claustrophobia)

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 160 subjects are anticipated, with the expectation that initial cognitive evaluations will exclude about 60 subjects. We intend to maintain and follow 100 subjects, 40 with non-dementia memory impairment (meeting criteria for amnestic MCI) and 40 with no cognitive impairment, and 20 with mild Alzheimer disease
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2009-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Clark, MD, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (1):
- Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark DG; Alzheimer Disease Neuroimaging Initiative. Residual vectors for Alzheimer disease diagnosis and prognostication. Brain Behav. 2011 Nov;1(2):142-52. doi: 10.1002/brb3.19. PMID 22399094
- [Result] Clark DG, Wadley VG, Kapur P, DeRamus TP, Singletary B, Nicholas AP, Blanton PD, Lokken K, Deshpande H, Marson D, Deutsch G. Lexical factors and cerebral regions influencing verbal fluency performance in MCI. Neuropsychologia. 2014 Feb;54:98-111. doi: 10.1016/j.neuropsychologia.2013.12.010. Epub 2013 Dec 30. PMID 24384308
- [Result] Clark DG, Kapur P, Geldmacher DS, Brockington JC, Harrell L, DeRamus TP, Blanton PD, Lokken K, Nicholas AP, Marson DC. Latent information in fluency lists predicts functional decline in persons at risk for Alzheimer disease. Cortex. 2014 Jun;55:202-18. doi: 10.1016/j.cortex.2013.12.013. Epub 2014 Jan 16. PMID 24556551

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All individuals underwent baseline MRI, cognitive, and functional assessment. Four individuals (2 cognitive impairment- non dementia (CIND), 1 intoxicated, 1 with non-AD dementia) determined not to fit into one of the study arms (MCI, mild AD, or cognitively normal) were not asked to return for follow up cognitive and functional assessment.
Groups:
- CIND: Individuals with cognitive impairment who did not meet criteria for MCI or dementia
- Intoxicated: Individuals who appeared to be intoxicated at baseline evaluation
- Non-AD Dementia: Other causes of dementia
Period: Overall Study
Arm/Group | Arm 1: Non-Dementia Memory Disorder | Arm 2: Control | Arm 3: Mild Alzheimer Disease | CIND | Intoxicated | Non-AD Dementia
Started | 23 | 40 | 11 | 2 | 1 | 1
Completed | 13 | 23 | 6 | 0 | 0 | 0
Not Completed | 10 | 17 | 5 | 2 | 1 | 1
Not completed — Physician Decision | 0 | 8 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of resources (hired rater) | 9 | 7 | 5 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Seventy-eight individuals underwent the baseline assessment, but four were removed from the analysis and were not asked to follow up because the consensus panel did not feel that they met criteria for any of the three arms (MCI, control, mild AD). This left 74 individuals at baseline who were eligible to continue in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Non-Dementia Memory Disorder | Arm 2: Control | Arm 3: Mild Alzheimer Disease | Total
Number analyzed (Participants) | 23 | 40 | 11 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.91 (7.63) | 65.08 (9.46) | 74.18 (6.29) | 68.55 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 23 | 3 | 30
  Male | 19 | 17 | 8 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 6 | 1 | 9
  White | 21 | 34 | 10 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Educational level [Mean (Standard Deviation); unit: years] | 14.9 (2.94) | 16.0 (2.39) | 14.8 (2.36) | 15.4 (2.6)
Verbal learning - 1st immediate list A [Mean (Standard Deviation); unit: words recalled] — Participants were read a list of 16 words and asked immediately to recite back as many words as they could remember.
  words recalled | 5.0 (1.7) | 6.4 (2.2) | 3.3 (1.4) | 5.4 (2.2)
Verbal learning - list B immediate recall [Mean (Standard Deviation); unit: words recalled] — After all 5 learning trials with list A, participants were read a second list of 16 words and asked immediately to recite back as many words as they could recall.
  words recalled | 4.5 (1.4) | 5.5 (2.2) | 2.7 (1.3) | 4.7 (2.0)
Verbal learning - total trials 1-5 [Mean (Standard Deviation); unit: words recalled] — Participants were read a list of 16 words five times in a row, each time being asked immediately to recite back as many words as they could recall. The sum of words recalled on the five attempts is reported here.
  words recalled | 35.9 (9.6) | 48.7 (10.0) | 23.0 (8.2) | 40.5 (13.2)
Verbal learning - long delay free recall [Mean (Standard Deviation); unit: words recalled] — After 30 minutes, participants were asked to recall words from list A (not from list B) that were presented during five previous exposure trials.
  words recalled | 5.8 (3.9) | 10.3 (3.5) | 1.6 (2.0) | 7.5 (4.6)
Verbal learning - long delay cued recall [Mean (Standard Deviation); unit: words recalled] — After attempting to spontaneously recall words from list A (following a 30 minute delay), participants were asked to recall all words they could recall within certain categories: animals, vegetables, articles of furniture, and ways of traveling (4 words in each category).
  words recalled | 7.3 (3.7) | 11.2 (3.2) | 3.3 (2.4) | 8.7 (4.3)
10/36 spatial recall - 1st trial [Mean (Standard Deviation); unit: positions recalled] — Participants were shown a 6 x 6 grid with black circles on 10 of the squares. After inspecting it for 10 seconds, they were given a blank grid and asked to place black checkers where the circles had been. This score is the number of checkers that were placed in actual locations of the circles.
  positions recalled | 4.3 (2.0) | 5.6 (2.0) | 4.0 (1.6) | 5.0 (2.0)
10/36 spatial recall - total [Mean (Standard Deviation); unit: positions recalled] — Participants were given three chances to memorize the positions of 10 black circles on a 6 x 6 grid. This score is the total number of correct responses over the three learning trials.
  positions recalled | 15.9 (5.0) | 20.2 (5.0) | 13.8 (3.0) | 17.9 (5.3)
10/36 spatial recall - delayed recall [Mean (Standard Deviation); unit: positions recalled] — After three exposures to a 6 x 6 grid with 10 black circles on it, participants were given a different task for 7 minutes and then asked to reproduce the pattern of circles by placing checkers on a blank grid. This score is the total number of correctly placed checkers.
  positions recalled | 5.2 (2.2) | 7.2 (2.4) | 5.4 (1.7) | 6.4 (2.4)
F-, A-, and S-words [Mean (Standard Deviation); unit: words generated] — Participants were given one minute each to generate as many words as possible that started with the letter F, the letter A, and the letter S. They were instructed not to use capitalized words, such as France, Friday, or Francheska. We report the sum of valid responses over the three tasks.
  words generated | 29.1 (14.5) | 36.4 (11.4) | 27.5 (14.0) | 32.5 (13.2)
Semantic fluency (7 categories) [Mean (Standard Deviation); unit: words generated] — Participants were given one minute to generate words fitting into 7 different semantic categories. We report the sum of valid responses over the 7 tasks. The categories were: animals, water creatures, tools, vehicles, fruits and vegetables, boats, and verbs.
  words generated | 74.6 (25.7) | 101.1 (23.3) | 61.5 (25.9) | 86.2 (28.5)
Trail Making Test - A [Mean (Standard Deviation); unit: seconds] — Participants were asked to draw a trial connecting labeled in circles in order. The labels consisted of the numbers from 1 to 25 and participants were told to start at 1 and finish at 25. We report the time in seconds for participants to complete the task.
  seconds | 45.4 (13.8) | 34.7 (11.4) | 77.0 (67.7) | 44.0 (30.1)
Trail Making Test - B [Mean (Standard Deviation); unit: seconds] — Participants were asked to draw a trial connecting circles in order according to the labels. The labels consisted of the numbers 1-13 and the letters A-M. Participants were told to alternate between numbers and letters (i.e., 1 - A - 2 - B - 3 - C, etc.) and were given a short practice form. We report the time taken to complete the task.
  seconds | 132.2 (64.4) | 78.8 (25.5) | 178.7 (79.2) | 110.8 (63.6)
Boston Naming Test - 30 item [Mean (Standard Deviation); unit: pictures named] — Participants were shown line drawings of objects and asked to name them. The test starts with highly familiar, high frequency words, such as 'bed,' and 'pencil,' and progresses to more difficult items, such as 'abacus' and 'octopus.' We report the number of correctly named items out of stimuli.
  pictures named | 25.6 (4.1) | 27.2 (2.2) | 21.6 (5.7) | 25.8 (4.0)
Pyramids and Palm Trees - pictures [Mean (Standard Deviation); unit: correct matches] — Participants were cued with a line drawing (e.g., a pyramid) and asked to decide which one of two other line drawings was most related to the cue. For the prototypical test item, the target and foil were, respectively, a palm tree and a pine tree. We report the number of correct items out of 51.
  correct matches | 49.4 (1.5) | 49.6 (1.4) | 46.4 (5.1) | 48.9 (2.6)
Pyramids and Palm Trees - words [Mean (Standard Deviation); unit: correct matches] — Participants were cued with a word (e.g., "pyramid") and asked to decide which one of two other words was most related to the cue. For the prototypical test item, the target and foil were, respectively, "palm tree" and "pine tree." We report the number of correct items out of 52.
  correct matches | 50.0 (1.8) | 50.4 (1.2) | 48.4 (4.9) | 49.9 (2.5)
Extended Mini-Mental State Exam [Mean (Standard Deviation); unit: points awarded for correct items] — The extended mini-mental state exam (xMMSE) is a 50-item test consisting of the 30 items from the standard MMSE, plus items that a give total of 20 additional possible points. The additional items are 5 points for an executive/working memory task, 2 points for naming, 6 points for delayed recall (with and without cues), 3 additional points for the visual construction, and 4 additional points for recalling the visual construction after a delay.
  points awarded for correct items | 44.2 (4.9) | 47.6 (2.5) | 36.5 (4.4) | 44.7 (5.2)
Financial Capacity Instrument - total [Mean (Standard Deviation); unit: points awarded for correct items] — The Financial Capacity Instrument is a test of financial knowledge and skills. We used items from five of the domains that have been previously reported: financial concepts (range 0-34), cash transactions (range 0-32), checkbook management (range 0-30), bank statement management (range 0-49), and bill payment (range 0-46). The number of points awarded for correct items depends on the estimated difficulty of the item. We report the sum of all points awarded across the five domains at the baseline evaluation (range 0-191), with higher scores representing greater financial capacity.
  points awarded for correct items | 151.8 (17.3) | 160.2 (8.3) | 127.1 (27.9) | 152.4 (19.0)

OUTCOME MEASURES:

1. Primary Outcome: FCI Score at Follow-up
Description: At each research visit, participants undertook 5 portions of the Financial Capacity Instrument (Domains 2, 3, 4b, 5, and 7). We report the total FCI score across the five domains tested, which has a range of possible scores from 0-191. Higher scores reflect greater capacity for understanding financial concepts and handling financial tasks.
Time Frame: Year 1, Year 2, Year 3
Population: Individuals completing at least one assessment following baseline
Measure: Mean (Standard Deviation); unit: points awarded for correct items
Arm/Group | Arm 1: Non-Dementia Memory Disorder | Arm 2: Control | Arm 3: Mild Alzheimer Disease
Number analyzed (Participants) | 10 | 22 | 6
points awarded for correct items
  Year 1 | 147.3 (19.7) | 164.0 (13.3) | 123.3 (43.1)
  Year 2 | 150.8 (9.0) | 179.0 (6.2) | 0 (0)
  Year 3 | 93 (0) | 163 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Potential adverse events were discussed at each research visit. For some patients, adverse events were detected through clinical interaction with the participants.
Arm/Group | Arm 1: Non-Dementia Memory Disorder | Arm 2: Control | Arm 3: Mild Alzheimer Disease | CIND | Intoxicated | Non-AD Dementia
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/40 | 0/11 | 0/2 | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 0/23 | 0/40 | 0/11 | 0/2 | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Non-Dementia Memory Disorder (N=23) | Arm 2: Control (N=40) | Arm 3: Mild Alzheimer Disease (N=11) | CIND (N=2) | Intoxicated (N=1) | Non-AD Dementia (N=1)
Death (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — This participant died from multi-organ failure within 3 months of the baseline evaluation.

LIMITATIONS AND CAVEATS:
This trial did not involve an intervention. Technical problems limited the analysis of the MRI scans. Lack of a designated rater for the study negatively impacted participant retention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes